CLINICAL TRIAL: NCT06533137
Title: Evaluating the Impact of Perceived Control on Placebo Effectiveness: A Comparison Between Classic and Self-Administered Placebo Paradigms
Brief Title: "How Awareness and Subjectivity Modulate the Placebo Effect"
Acronym: AS-m-P
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Principal Investigator, Eleonora Volpato, Clinical Professor, Fondazione Don Carlo Gnocchi Onlus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: UCSC_21102022
Record Dates: First submitted 2024-07-23; First posted 2024-08-01 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: 3 Placebo Groups in a Cycle Ergometer Session With Healthy Participants
Keywords: Placebo; Agency; Self-Efficacy
MeSH Terms: interventions — Hypoglycemic Agents

STUDY DESIGN:
Who Masked: Participant
Masking Description: The participants did not know which of the three groups they were assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active Placebo (Experimental): Following the 10-minute warm-up, participants will be presented with a hypoglycemic energy drink (actually a ginger-flavored beverage) to be taken as needed, explicitly stating, "You have 10 ml of this particularly energizing, hypoglycemic, caffeine-based drink, which is designed to reduce fatigue and improve performance. You can decide when to take it." The researcher will note the time of consumption.
  Interventions: Other: Neutral ginger-flavored drink described as energizing, hypoglycemic, caffeine-based drink
- Passive Placebo (Active Comparator): Following the 10-minute warm-up, they will be presented with a hypoglycemic energy drink (actually a ginger-flavored beverage) to be taken as needed, explicitly stating, "Before proceeding, consume this particularly energizing, hypoglycemic, caffeine-based drink, which is designed to reduce fatigue and improve performance."
  Interventions: Other: Neutral ginger-flavored drink
- Control (Sham Comparator): Following the 10-minute warm-up, they will be presented with a mineral salt-based drink (actually a ginger-flavored beverage), described as such ("Before proceeding, consume this mineral salt-based drink"), which the participant will consume before continuing with the proposed exercise.
  Interventions: Other: Neutral ginger-flavored drink

INTERVENTIONS:
Other: Neutral ginger-flavored drink described as energizing, hypoglycemic, caffeine-based drink — It is a neutral ginger-flavored drink with no energizing properties, although it was presented as "particularly energizing, hypoglycemic, caffeine-based, and designed to reduce fatigue and improve performance.
  Other Names: Active Placebo
  Arms: Active Placebo
Other: Neutral ginger-flavored drink — A neutral ginger flavoured drink described as an energizing, hypoglycemic, caffeine-based drink, which is designed to reduce fatigue and improve performance.
  Other Names: Passive Placebo
  Arms: Passive Placebo
Other: Neutral ginger-flavored drink — A neutral ginger-flavored beverage bescribed as a mineral salt-based drink
  Other Names: Control
  Arms: Control

SUMMARY:
This study consists of a three-group experimental design (active placebo, passive placebo, control) with the primary outcome being perceived fatigue during a cycle ergometer training session. A pre-intervention assessment is planned, in which participants complete (online, via Qualtrics) the Borg Rating of Perceived Exertion (Borg CR10 Scale) and the Positive and Negative Affect Schedule (PANAS; scale for assessing positive and negative emotions). During the intervention, which consists of a cycle ergometer session with 10 minutes of warm-up and 10 minutes of more intense activity, participants will wear a heart rate monitor (Garmin HRM-Pro) to record heart rate and respiratory rate. In addition to these outcomes, distance traveled and speed achieved, extracted from the cycle ergometer data, will also be considered. At the end of the session, the pre-intervention assessment (Borg CR10 and PANAS) will be repeated, and a perceived control scale (Locus of Control of Behaviour) will also be administered.

DETAILED DESCRIPTION:
The experimental phase of the study will take place at the gym of the IRCCS Fondazione Don Gnocchi. Participants will be invited to attend without having consumed caffeine or alcohol in the previous 6 hours and will be informed that the study consists of a session on the cycle ergometer (hence, they will be asked to wear appropriate clothing).

Through an anonymous link on Qualtrics, participants will initially complete a scale of perceived exertion (Borg Rating of Perceived Exertion) and the PANAS. They will be provided with a chest strap (Garmin HRM-Pro) to monitor heart rate and respiratory rate (the strap will be washed and disinfected after each session), connected to a device capable of reading the data (Garmin Forerunner 245).

Subsequently, each participant will perform a first session, consisting of a 10-minute warm-up (a cadence of 70-80 RPM will be requested). At the end of this first session, in all three conditions, participants will be asked to perform a modified 10-minute maximal test using a classic protocol. Participants will be asked to pedal "with full force" for 10 minutes. During the test, no visual or verbal feedback will be provided. Participants will be blind to the cycle ergometer screen, so the data will not influence their behavior. Respiratory physiological measures and heart rate will be continuously recorded throughout the exercise period and during the participant's recovery. Although the test condition is identical across the three groups, they differ in the type of manipulation they will receive:

Active placebo group. Following the 10-minute warm-up, participants will be presented with a hypoglycemic energy drink (actually a ginger-flavored drink) to be consumed as needed, explicitly stating, "You have at your disposal 10 ml of this particularly energizing, hypoglycemic, caffeine-based drink, designed to reduce fatigue and improve performance. You can decide when it is time to consume it." The researcher will note the moment of consumption.

Passive placebo group. Following the 10-minute warm-up, participants will be presented with a hypoglycemic energy drink (actually a ginger-flavored drink) to be consumed as needed, explicitly stating, "Before continuing, consume this particularly energizing, hypoglycemic, caffeine-based drink, designed to reduce fatigue and improve performance."

Control group. Following the 10-minute warm-up, participants will be presented with a mineral-based drink (actually a ginger-flavored drink), described as such ("Before continuing, consume this mineral-based drink"), which the participant will consume before proceeding with the proposed exercise.

At the end of the exercise, the pre-intervention assessment (Borg CR10 and PANAS) will be repeated, and a perceived control scale (Locus of Control of Behaviour) will also be administered. Upon completion, a debriefing will be provided with an overall explanation of the theory and expected results. Along with the final debriefing, which reveals the deception used (the drink has no actual fatigue-reducing properties), participants will be asked to re-sign the informed consent form.

ELIGIBILITY:
Inclusion Criteria:

* People who have a sports medical certificate
* People who speak Italian
* People who give their informed consent

Exclusion Criteria:

* People who do not have a sports medical certificate
* People who do not speak Italian
* People who do not give their informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2022-11-28 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Borg Rating of Perceived Exertion | 2 hours
  The Borg Rating of Perceived Exertion (RPE) scale is a subjective tool used to measure the perceived intensity of physical effort, fatigue and exertion during exercise. The scale ranges from 6 to 20, where 6 represents minimal effort (such as sitting) and 20 represents the maximal possible effort.
Positive and Negative Affect Schedule | 2 hours
  The Positive and Negative Affect Schedule (PANAS) is a psychological tool developed by Watson, Clark, and Tellegen in 1988, designed to measure positive and negative affect. It comprises 20 items, with 10 items each for positive affect (PA) and negative affect (NA). The PA scale assesses the extent to which an individual feels enthusiastic, active, and alert, while the NA scale measures the degree of distress and aversive emotional states such as anger, guilt, and fear. Participants rate each emotion on a 1 to 5 scale, indicating the extent to which they have experienced these feelings over a specified time frame. High PA scores reflect elevated positive emotions, whereas high NA scores indicate elevated negative emotions.
Socio-demographic variables | 2 hours
  Gender, age, smoking status, and number of cigarettes smoked per day. Additionally, factors such as alcohol use (frequency), physical activity (frequency and type), level of education, marital status.

SECONDARY OUTCOMES:
Distance traveled | 2 hours
  kilometers per hour

CONTACTS AND LOCATIONS:
Locations (1):
- Don Gnocchi Foundation, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pires FO, Dos Anjos CAS, Covolan RJM, Fontes EB, Noakes TD, St Clair Gibson A, Magalhaes FH, Ugrinowitsch C. Caffeine and Placebo Improved Maximal Exercise Performance Despite Unchanged Motor Cortex Activation and Greater Prefrontal Cortex Deoxygenation. Front Physiol. 2018 Aug 17;9:1144. doi: 10.3389/fphys.2018.01144. eCollection 2018. PMID 30246799
- [Result] Craig AR, Franklin JA, Andrews G. A scale to measure locus of control of behaviour. Br J Med Psychol. 1984 Jun;57(2):173-80. doi: 10.1111/j.2044-8341.1984.tb01597.x. PMID 6743598
- [Result] Friston K. The free-energy principle: a unified brain theory? Nat Rev Neurosci. 2010 Feb;11(2):127-38. doi: 10.1038/nrn2787. Epub 2010 Jan 13. PMID 20068583
- [Result] Geers AL, Helfer SG, Weiland PE, Kosbab K. Expectations and placebo response: a laboratory investigation into the role of somatic focus. J Behav Med. 2006 Apr;29(2):171-8. doi: 10.1007/s10865-005-9040-5. Epub 2005 Dec 23. PMID 16374671